CLINICAL TRIAL: NCT04554368
Title: A Novel Score to Predict Risk of Symptomatic Intracerebral Hemorrhage After Stroke Thrombectomy: Derivation, Validation and Comparison With Other Scores
Brief Title: A Novel Score to Predict Risk of Symptomatic Intracerebral Hemorrhage
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yueqi Zhu, Clinical Professor, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Other Study IDs: Henan-PRIH score
Record Dates: First submitted 2020-09-13; First posted 2020-09-18 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Intracerebral Hemorrhage; Thrombectomy; Stroke
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IA-CEFDCT group: 95 patients who underwent IA-CEFDCT and MT for acute anterior stroke.
  Interventions: Procedure: intra-arterial contrast enhanced Flat Detector CT

INTERVENTIONS:
Procedure: intra-arterial contrast enhanced Flat Detector CT — After femoral artery puncture, FDCT scan (if necessary) and IA-CEFDCT scan were performed on a single flat-detector angiography system (Allura Xper FD20, Philips Medical systems, Best, the Netherlands), respectively. FDCT was acquired with the following acquisition parameters: 20s rotation, 220° rotation, 617 single frames at a frame rate of 30/s, 48cm detector field of view, 1024 acquisition matrix. Images were reconstructed using a soft-tissue kernel with an isotropic voxel size of 0.9 × 0.9 × 0.9 mm on a dedicated workstation for FPCT data (XperCT Dual 3.2.0). For image analysis, these isotropic FDCT data were viewed in the axial plane with 5 mm slice thickness.

SUMMARY:
This study sought to develop and validate a new risk stratification score (Henan predicting the risk of intracerebral hemorrhage score, Henan-PRIHS) based on intra-arterial contrast enhanced Flat Detector CT (IA-CEFDCT) to predict symptomatic intra-cerebral hemorrhage (sICH) after stroke thrombectomy.

DETAILED DESCRIPTION:
The Henan-PRIHS was developed from 95 patients who underwent IA-CEFDCT and MT for acute anterior stroke. Patients were classified as having one of three grades according to the presence of contrast filling within the occluded vascular territory. Grade 0 was normal or less contrast filling in affected hemisphere, grade 1 and 2 were small and medium-large area without contrast filling, respectively. The Youden index was used to determine the optimum no contrast filling area cutoff for defining grade 1 and 2. The score was subsequently validated in a different population of 208 patients and compared with three established scores.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years,
2. occlusion of internal carotid artery and/or middle cerebral artery (MCA) M1 or M2 segments confirmed by CTA or MRA or DSA,
3. baseline National Institutes of Health Stroke Scale (NIHSS) score ≥ 4 points,
4. MT was performed within 16 hours from stroke onset,
5. baseline CT scan and IA-CEFDCT scan must be performed; 24 hours post-treatment CT scan was done and when the patient's neurological state had deteriorated.

Exclusion Criteria:

1. bilateral infarcts,
2. history of hemorrhagic stroke,
3. post-procedure ICH (including SAH) due to iatrogenic complications,
4. missing clinical and demographic data,
5. poor-quality IA-CEFDCT scans (i.e., motion artifact) that limited accurate identification of the region of interest. Bridge treatment (combined intravenous thrombolysis with MT) was not excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute anterior circulation stroke
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Henan predicting the risk of intracerebral hemorrhage score | 5 days
  Grade 0 was normal or less contrast filling in affected hemisphere, grade 1 and 2 were small and medium-large area without contrast filling, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai 6th People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made avaliable